CLINICAL TRIAL: NCT01340053
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Assess the Safety and Efficacy of RDX5791 for the Treatment of Constipation-Predominant Irritable Bowel Syndrome (IBS-C)
Brief Title: A Study to Evaluate the Safety and Efficacy of RDX5791 for the Treatment of Constipation Predominant Irritable Bowel Syndrome (IBS-C)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ardelyx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RDX5791-201
Record Dates: First submitted 2011-04-20; First posted 2011-04-22 (Estimated); Results first posted 2019-10-15 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-09

CONDITIONS: Constipation Predominant Irritable Bowel Syndrome
MeSH Terms: interventions — tenapanor

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Capsule that is identical in size and color to other treatments
  Interventions: Drug: RDX5791
- Low Dose (Experimental): 10 mg capsule of tenapanor
  Interventions: Drug: RDX5791
- Mid Dose (Experimental): 30 mg capsule of tenapanor
  Interventions: Drug: RDX5791
- High Dose (Experimental): 100 mg capsule of tenapanor
  Interventions: Drug: RDX5791

INTERVENTIONS:
Drug: RDX5791 — Capsule, QD

SUMMARY:
This is a multi-center, Phase 2, randomized, double-blind, placebo controlled study of RDX5791 in subjects with IBS-C. Patients who are 18 to 75 years old, meeting the definition of IBS-C as defined by the Rome III Criteria for the Diagnosis of IBS will undergo a battery of screening procedures to determine eligibility for the trial.

The study will consist of a 2-week treatment-free screening period, a 4-week blinded treatment period, and a 2-week treatment-free follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Subject meets Rome III criteria for IBS-C
* If > 50 years old, colonoscopy evaluation within 10 years
* All ages, negative colonoscopy if any "warning symptoms"
* Active disease during 2-week screening period
* Compliant with IVRS

Exclusion Criteria:

* Subjects has IBS-D, IBS-M or un-subtyped IBS according to Rome III criteria
* Diagnosis or treatment of any clinically symptomatic biochemical or structural abnormality of the GI tract
* Use of medications that are known to affect stool consistency
* Subject has any protocol-excluded or clinically significant medical or surgical history that could confound the study assessments or prevent completion of study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2011-05; Primary Completion 2011-12 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David P Rosenbaum, Ph.D., Study Chair — Ardelyx
Locations (16):
- United States (16):
  - Ardelyx Investigational Site, San Diego, California
  - Ardelyx Investigational Site, Jupiter, Florida
  - Ardelyx Investigational Site, Pinellas Park, Florida
  - Ardelyx Investigational Site, Rockford, Illinois
  - Ardelyx Investigational Site, Mission, Kansas
  - Ardelyx Investigational Site, Monroe, Louisiana
  - Ardelyx Investigational Site, Annapolis, Maryland
  - Ardelyx Investigational Site, Chesterfield, Michigan
  - Ardelyx Investigational Site, St Louis, Missouri
  - Ardelyx Investigational Site, Brooklyn, New York
  - Ardelyx Investigational Site, Greensboro, North Carolina
  - Ardelyx Investigational Site, Oklahoma City, Oklahoma
  - Ardelyx Investigational Site, Simpsonville, South Carolina
  - Ardelyx Investigational Site, Bristol, Tennessee
  - Ardelyx Investigational Site, Ogden, Utah
  - Ardelyx Investigational Site, Lynchburg, Virginia

REFERENCES:
- See also: Related Info — http://www.ardelyx.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo: Capsule, QD
- 10mg; 30 mg; 100 mg: RDX5791: Capsule, QD
Period: Overall Study
Arm/Group | Placebo | 10mg | 30 mg | 100 mg
Started | 47 | 46 | 47 | 46
Completed | 43 | 44 | 43 | 43
Not Completed | 4 | 2 | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Low Dose | Mid Dose | High Dose | Total
Number analyzed (Participants) | 47 | 46 | 47 | 46 | 186
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.9 (11.97) | 44.4 (14.15) | 46.5 (9.49) | 43.5 (12.31) | 45.6 (12.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 42 | 39 | 37 | 157
  Male | 8 | 4 | 8 | 9 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 6 | 5 | 8 | 22
  Not Hispanic or Latino | 44 | 40 | 42 | 38 | 164
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 2 | 0 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 12 | 5 | 9 | 10 | 36
  White | 34 | 39 | 38 | 36 | 147
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.02 (5.56) | 27.40 (6.97) | 28.58 (6.10) | 28.10 (4.14) | 28.03 (5.74)

OUTCOME MEASURES:

1. Primary Outcome: Complete Spontaneous Bowel Movement (CSBM) Frequency Change From Baseline
Description: Patients complete a phone diary daily. They are asked "how many bowel movements have you had today?" they are then asked for each spontaneous bowel movement (unaided with laxative use) wether there was its was a complete evacuation. if it was then it is a complete spontaneous bowel movement. All CSBMs are added and adjusted for a mean compete sponteneous bowel movement.
Time Frame: Baseline and Week 4
Population: All patients randomized who received at least one dose of drug
Measure: Mean (Standard Deviation); unit: number of bowel movements/week
Arm/Group | Placebo | Low Dose | Mid Dose | High Dose
Number analyzed (Participants) | 47 | 45 | 47 | 46
number of bowel movements/week | 1.01 (2.03) | 1.50 (2.09) | 1.54 (2.10) | 1.57 (2.50)

2. Secondary Outcome: Spontaneous Bowel Movement (SBM) Frequency Change From Baseline
Time Frame: baseline and week 4
Measure: Mean (Standard Deviation); unit: change in number of bowel movements
Arm/Group | Placebo | Low Dose | Mid Dose | High Dose
Number analyzed (Participants) | 47 | 45 | 47 | 46
change in number of bowel movements | 1.58 (2.51) | 2.37 (2.27) | 2.97 (3.13) | 2.81 (3.14)

ADVERSE EVENTS:
Arm/Group | Placebo | Low Dose | Mid Dose | High Dose
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/46 | 0/47 | 0/46
Serious Adverse Events (participants affected / at risk) | 0/47 | 2/46 | 0/47 | 0/46
Other Adverse Events (participants affected / at risk) | 0/47 | 0/46 | 0/47 | 0/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=47) | Low Dose (N=46) | Mid Dose (N=47) | High Dose (N=46)
cholecystitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
appendicitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publications must be reviewed and approved by sponsor